CLINICAL TRIAL: NCT01152437
Title: An Open Label, Partially Randomised Phase II Study to Investigate the Efficacy and Safety of BIBW 2992 in Patients With Metastatic Colorectal Cancer Who Never Received Prior Anti-EGFR (Epidermal Growth Factor Receptor) Treatment
Brief Title: A Study of BIBW 2992 (Afatinib) in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.74; 2009-011996-59 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Afatinib; Cetuximab

ARMS (2):
- BIBW 2992 (Experimental): Patients receive BIBW 2992 tablets once daily
  Interventions: Drug: BIBW 2992
- Cetuximab (Active Comparator): Patients receive cetuximab intravenously once a week, every week
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: BIBW 2992 — Patients receive BIBW 2992 tablets once daily, and can reduce dose for adverse event management
  Arms: BIBW 2992
Drug: Cetuximab — Patients receive cetuximab intravenously, once a week, every week
  Arms: Cetuximab

SUMMARY:
This Phase II study is open to patients with metastatic colorectal cancer who have tried but failed chemotherapy regimens containing oxaliplatin and irinotecan. Patients must not have received anti-EGFR (Epidermal Growth Factor Receptor) treatment (for example, cetuximab, panitumumab) in the past. Patients with wild-type KRAS (v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog) colorectal cancer will be randomised to receive either BIBW 2992 or cetuximab. Patients with KRAS mutated colorectal cancer will not be randomised, but will all receive BIBW 2992. The main objectives of the study are: to compare the effectiveness of BIBW 2992 with that of cetuximab in patients with KRAS wild type cancer, and to assess the effectiveness of BIBW 2992 in patients with KRAS mutated cancer.

ELIGIBILITY:
Inclusion criteria:

1. Patients with metastatic colorectal cancer who have failed both oxaliplatin- and irinotecan-based regimens
2. Tumour sample available for KRAS (v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog) mutation testing and other biomarker analyses.

Exclusion criteria:

1. Prior treatment with Epidermal Growth Factor Receptor (EGFR) targeting small molecules or antibodies.
2. Biological treatment (including Bevacizumab or any other antiangiogenic agents) during the trial is not allowed.
3. Known pre-existing interstitial lung disease.
4. Planned major surgical procedures during the trial period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (13):
- United Kingdom (13):
  - 1200.74.44001 Boehringer Ingelheim Investigational Site, Bournemouth
  - 1200.74.44005 Boehringer Ingelheim Investigational Site, Bristol
  - 1200.74.44006 Boehringer Ingelheim Investigational Site, Cambridge
  - 1200.74.44003 Boehringer Ingelheim Investigational Site, Glasgow
  - 1200.74.44009 Boehringer Ingelheim Investigational Site, London
  - 1200.74.44012 Boehringer Ingelheim Investigational Site, Manchester
  - 1200.74.44007 Boehringer Ingelheim Investigational Site, Northwood
  - 1200.74.44013 Boehringer Ingelheim Investigational Site, Nottingham
  - 1200.74.44011 Boehringer Ingelheim Investigational Site, Poole
  - 1200.74.44010 Boehringer Ingelheim Investigational Site, Sheffield
  - 1200.74.44008 Boehringer Ingelheim Investigational Site, Southampton
  - 1200.74.44004 Boehringer Ingelheim Investigational Site, Sutton, Surrey
  - 1200.74.44002 Boehringer Ingelheim Investigational Site, Truro

RESULTS

PARTICIPANT FLOW:
Groups:
- Afatinib (Wild-type): Afatinib tablets once daily in patients with KRAS (v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog) wild-type metastatic colorectal cancer. Patients started on 40 mg and then increased to 50 mg after 4 weeks if well tolerated.
- Cetuximab (Wild-type): Cetuximab 400 mg/m² on Day 1 and then 250mg/m² once a week, every week, intravenous (i.v.) in patients with KRAS wild-type metastatic colorectal cancer.
- Afatinib (Mutated): Afatinib tablets once daily in patients with KRAS mutated metastatic colorectal cancer. Patients started on 40 mg and then increased to 50 mg after 4 weeks if well tolerated.
Period: Overall Study
Arm/Group | Afatinib (Wild-type) | Cetuximab (Wild-type) | Afatinib (Mutated)
Started | 36 (randomised) | 15 (randomised) | 43 (entered)
Completed | 0 | 0 | 0
Not Completed | 36 | 15 | 43
Not completed — Other Adverse Event | 8 | 1 | 7
Not completed — Not treated | 0 | 1 | 2
Not completed — Progressive disease | 27 | 13 | 32
Not completed — Refusal to continue taking trial medicat | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Treated set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib (Wild-type) | Cetuximab (Wild-type) | Afatinib (Mutated) | Total
Number analyzed (Participants) | 36 | 14 | 41 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.4) | 62.6 (7.7) | 60.0 (11.9) | 61.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 22 | 36
  Male | 27 | 9 | 19 | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response: complete response (CR) or partial response (PR) according to RECIST (version 1.1) without confirmation criteria applied.
Time Frame: Baseline till progression or death, whichever came first, assessed up to 23 months
Population: Randomised set. Primary endpoint for the population of patients with KRAS wildtype tumours.
Measure: Number; unit: Percentage of Participants
Arm/Group | Afatinib (Wild-type) | Cetuximab (Wild-type)
Number analyzed (Participants) | 36 | 15
Percentage of Participants | 3 | 20
Statistical Analysis 1: Comparison: Afatinib (Wild-type) vs Cetuximab (Wild-type); Null hypothesis is that the objective response rate (ORR) in KRAS wild-type patients treated with afatinib is less than or equal to the ORR in KRAS wild-type patients treated with cetuximab. Sample size is based on a 'pick the winner' approach assuming ORR for cetuximab of 12%, undesirable ORR for afatinib of 11% and desirable ORR for afatinib of 16%. As per 'pick the winner' approach, afatinib would be considered 'the winner' if the ORR for afatinib was greater than the ORR for cetuximab; Test type: Superiority or Other; p = 0.0735, Regression, Logistic — The statistical analysis is descriptive and exploratory in nature and performed only to provide a statistical framework from which to view the results and plan further studies; Wald Chi-square test and Confidence Interval from logistic regression stratified by number of lines of palliative chemotherapy; Odds Ratio (OR) = 0.122, 90% CI 2-sided [0.018 to 0.844]

2. Primary Outcome: Percentage of Participants With Disease Control (DC)
Description: Percentage of participants with objective response or stable disease (SD) as determined by RECIST (version 1.1) with confirmation criteria applied.
Time Frame: Baseline till progression or death, whichever came first, assessed up to 23 months
Population: Treated Set. Primary endpoint for the population of patients with KRAS mutated tumours.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Afatinib (Mutated)
Number analyzed (Participants) | 41
Percentage of Participants | 12 [4.9 to 23.9]
Statistical Analysis 1: Comparison: Afatinib (Mutated); Null hypothesis is that the disease control rate is 10% in patients with KRAS mutation. Sample size calculation based on a 2-sided exact binomial test at 10% significance level to distinguish between the historical disease control rate of 10% and a desirable disease control rate for afatinib of 25%; Test type: Superiority or Other; p = 0.6394, Exact binomial test — [p-value comment as in outcome 1, analysis 1]; Percentage of participants = 12, 90% CI 2-sided [4.9 to 23.9]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS time is defined as time from randomisation (wild-type group) or start of treatment (mutated group) to tumor progression evaluated according to RECIST (version 1.1) or death whichever occurs earlier. Median and confidence interval estimated using product-limit Kaplan-Meier method.
Time Frame: Baseline till progression or death, whichever came first, assessed up to 23 months
Population: Randomised set for wild-type group and treated set for mutated group.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Afatinib (Wild-type) | Cetuximab (Wild-type) | Afatinib (Mutated)
Number analyzed (Participants) | 36 | 15 | 41
Days | 46.0 [43.0 to 49.0] | 144.5 [24.0 to 233.0] | 41.0 [39.0 to 46.0]

4. Secondary Outcome: Overall Survival (OS) Time
Description: OS time is defined as time from the date of randomisation (wild-type group) or date of start of treatment (mutated group) to the date of death. Median and confidence interval estimated using product-limit Kaplan-Meier method.
Time Frame: Baseline till death, assessed up to 23 months
Population: Randomised set for wild-type group and treated set for mutated group.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Afatinib (Wild-type) | Cetuximab (Wild-type) | Afatinib (Mutated)
Number analyzed (Participants) | 36 | 15 | 41
Days | 355.0 [211.0 to 449.0] | NA [204.0 to NA] — NA - This was not calculable due to the low number of deaths observed in this group. | 173.0 [106.0 to 214.0]

5. Secondary Outcome: Pre-dose Concentration of Afatinib in Plasma at Steady State on Day 8 (Cpre,ss,8)
Description: Cpre,ss,8 represents the pre-dose concentration of afatinib in plasma at steady state on day 8.
Time Frame: day 8
Population: Randomised set for wild-type group and treated set for mutated group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib (Wild-type) | Afatinib (Mutated)
Number analyzed (Participants) | 28 | 24
ng/mL | 16.6 (80.3) [211.0 to 449.0] | 21.4 (91.0) [106.0 to 214.0]

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Arm/Group | Afatinib (Wild-type) | Cetuximab (Wild-type) | Afatinib (Mutated)
Serious Adverse Events (participants affected / at risk) | 15/36 | 5/14 | 18/41
Other Adverse Events (participants affected / at risk) | 35/36 | 14/14 | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (Wild-type) (N=36) | Cetuximab (Wild-type) (N=14) | Afatinib (Mutated) (N=41)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 4
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 5
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1 | 3
Condition aggravated (General disorders) | 1 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 4
Fatigue (General disorders) | 1 | 1 | 1
Malaise (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 2 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 1
Ureteritis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood calcium increased (Investigations) | 0 | 0 | 1
Quality of life decreased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 2 | 0 | 0
Speech disorder (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (Wild-type) (N=36) | Cetuximab (Wild-type) (N=14) | Afatinib (Mutated) (N=41)
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 2 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0
Scintillating scotoma (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 7
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 10 | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 25 | 4 | 25
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 3
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 12 | 3 | 17
Oral pain (Gastrointestinal disorders) | 7 | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 4
Rectal tenesmus (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 6 | 3 | 8
Vomiting (Gastrointestinal disorders) | 6 | 2 | 14
Chills (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 12 | 3 | 15
Influenza like illness (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 3 | 1 | 3
Oedema peripheral (General disorders) | 2 | 2 | 5
Pain (General disorders) | 2 | 1 | 3
Pyrexia (General disorders) | 0 | 2 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0
Oral candidiasis (Infections and infestations) | 2 | 0 | 3
Oral herpes (Infections and infestations) | 1 | 1 | 0
Paronychia (Infections and infestations) | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 4 | 3 | 6
Weight decreased (Investigations) | 2 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 11 | 6 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 5 | 0 | 4
Headache (Nervous system disorders) | 2 | 4 | 4
Lethargy (Nervous system disorders) | 2 | 3 | 4
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 1 | 2
Proteinuria (Renal and urinary disorders) | 3 | 1 | 4
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 | 2 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 4
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 19 | 10 | 25
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 4
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.